CLINICAL TRIAL: NCT03209193
Title: Effect of Anesthetics on Microcirculation in Patients Undergoing Off-pump Coronary Artery Bypass Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Youn Joung Cho, MD, Clinical Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OPCAB_SEVO vs DES
Record Dates: First submitted 2017-07-03; First posted 2017-07-06 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Microcirculation; Anesthetic Complication Spinal
Keywords: off-pump coronary artery bypass; sevoflurane; desflurane; tissue oxygen saturation
MeSH Terms: interventions — Sevoflurane; Desflurane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sevoflurane (Experimental): Sevoflurane (2 vol%) use as a maintenance volatile anesthetic drug during the surgery
  Interventions: Drug: Sevoflurane
- Desflurane (Experimental): Desflurane (6 vol%) use as a maintenance volatile anesthetic drug during the surgery
  Interventions: Drug: Desflurane

INTERVENTIONS:
Drug: Sevoflurane — Sevoflurane use as main anesthetic drug during the surgery
  Arms: Sevoflurane
Drug: Desflurane — Desflurane use as main anesthetic drug during the surgery
  Arms: Desflurane

SUMMARY:
Volatile anesthetics, such as sevoflurane and desflurane, are commonly used in patients undergoing cardiac surgeries including off-pump coronary artery bypass. However, the effect of volatile anesthetics on microcirculation in patients undergoing off-pump coronary artery bypass has not been well conducted.

DETAILED DESCRIPTION:
This is a prospective randomized clinical trial investigating the effect of sevoflurane vs. desflurane on tissue microcirculation in patients undergoing off-pump coronary artery bypass surgery. Eligible patients are going to be randomized to receive sevoflurane or desflurane, as a maintenance anesthetic, during the surgery. Tissue oxygen saturation and microcirculatory changes, such as an occlusion and recovery slope, during vascular occlusion test will be recorded during the surgery. The primary end point of the study is the difference in tissue oxygen saturation between the groups.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for off-pump coronary artery bypass surgery

Exclusion Criteria:

* any deformity or vascular abnormalities on upper arms
* cannot receive sevoflurane or desflurane for any reason (muscular diseases, etc)
* uncontrolled diabetes
* peripheral vascular disease
* severe renal dysfunction (end-stage renal disease)
* refuse to enroll
* pregnant

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2017-07-04 (Actual); Primary Completion 2019-11-07 (Actual); Study Completion 2019-11-07 (Actual)

PRIMARY OUTCOMES:
Tissue oxygen saturation measured at thenar eminence by Hutchinson(R) tissue oximeter during off-pump coronary artery bypass surgery | Before induction of anesthesia to the end of the surgery, an average 8 hours
  Tissue oxygen saturation measured at thenar eminence by tissue oximeter during surgery in patients receiving sevoflurane or desflurane

CONTACTS AND LOCATIONS:
Overall Officials: Youn Joung Cho, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cho YJ, Yoo SJ, Nam K, Bae JY, Lee SH, Jeon Y. Effects of anesthetics on microvascular reactivity measured by vascular occlusion tests during off-pump coronary artery bypass surgery: a randomized controlled trial. J Clin Monit Comput. 2021 Oct;35(5):1219-1228. doi: 10.1007/s10877-020-00587-8. Epub 2020 Sep 11. PMID 32915370